CLINICAL TRIAL: NCT04008953
Title: Intravascular Volume Assessment Using Ultrasonography in Pediatrics Renal Transplant: A Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fatma Alzahraa Mohamed Ibrahim Hassan Haggag (Other)
Responsible Party: Sponsor-Investigator, Fatma Alzahraa Mohamed Ibrahim Hassan Haggag, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 2008@123
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Failure
Keywords: volume assessment
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sixteen patients having end stage renal disease: Intravascular volume assessment in 16 pediatric patients under going renal transplant surgery using ultrasonography, CVP and echocardiography
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — Intravascular volume assessment using ultrasonography, CVP and echocardiography

SUMMARY:
This study is designed for volume assessment in pediatrics during major surgery using non-invasive tools as ultrasonography without the need of invasive techniques avoiding its complications and as a guide for fluid therapy needed for maintaining adequate hemodynamics

DETAILED DESCRIPTION:
Intravascular volume assessment during surgery is important for maintaining adequate hemodynamics. Methods approved for volume assessment include the use of echocardiography to measure left ventricular end diastolic area (LVEDA), central venous pressure (CVP) and pulmonary artery diastolic pressure (PAD). LVEDA is considered the good predictor for volume status assessment. CVP and PAD are invasive can potentially subject the patient to complications. Recently study performed an ultrasound assessment of the internal jugular vein (IJV) as a useful means of volume status assessment intraoperative under general anesthesia. In the pediatric population, only few studies are carried out to assess the use of ultrasound for intravascular volume assessment. This study will evaluate use of Ultrasonography of IJV in volume assessment in pediatrics will undergo renal transplant surgery and correlate IJV diameter, cross sectional area to CVP and LVEDA.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with end stage renal disease
* Weight between: 12 to 30 kg

Exclusion Criteria:

* Infection at the site of CVP or generalized infection.
* IJV thrombosis

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sixteen consecutive pediatric patients having end stage renal disease scheduled for living related donor renal transplant surgery
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Internal jugular vein diameter, cross sectional area and left ventricular end-diastolic area | 3months
  Correlation of IJV diameter and cross sectional area to LVEDA.

SECONDARY OUTCOMES:
Internal jugular vein diameter, cross sectional area and central venous pressure | 3months
  Correlation of IJV diameter and cross sectional area to CVP.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Soaida, Study Director — Departement of Anesthesia Kasr Alainy Medical School Cairo University

IPD SHARING:
Plan to Share IPD: Undecided